CLINICAL TRIAL: NCT06433414
Title: Preventing Medication Complications During AcUte Illness Through Symptom Evaluation and Sick Day Guidance Mobile Application (PAUSE)
Brief Title: PAUSE: Sick Day Medication Management Mobile App Study
Acronym: PAUSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro000140652
Record Dates: First submitted 2024-05-13; First posted 2024-05-29 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Chronic Condition; Adverse Event
Keywords: chronic condition; medication safety; sick day medication guidance
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants receiving usual care will only receive the SDMG patient handout from their community pharmacist. This handout has been adapted from the Diabetes Canada "How to Stay Safe When You Are Sick" SDMG patient resource as well as the results of a modified Delphi study conducted by the research team to achieve consensus among 25 international clinicians on recommendations for SDMG for people with diabetes, kidney, or cardiovascular disease. This handout will be reviewed and refined with input from people with lived experience with the chronic conditions of interest prior to the study and is intended to provide guidance on how to self-manage medications during a sick day event.
- PAUSE App Intervention (Experimental): Participants will receive enhanced care through onboarding and accessing the PAUSE App via the PC Health app to provide continuity of care electronically through a personalized eHealth mobile application, as well as the SDMG patient resource handout. The PAUSE App provides the same guidance as the SDMG handout, but uses algorithms tailored to identify and provide guidance specific to users' symptoms and current medications.
  Interventions: Other: PAUSE App

INTERVENTIONS:
Other: PAUSE App — Participants receiving the intervention will receive access to the PAUSE App, a self-management tool for SDMG intended for patients to use during an acute illness. The app asks users a series of questions regarding signs and symptoms that identify a qualifying sick day illness, and screens for 'red flags' that would require emergency, or HCP or urgent care referral, and help patients identify which of their medications they should temporarily withhold or adjusted, tailored to a patients' current medication list. This aims to provide patients with interactive support for managing medication during a sick day event. As part of the intervention, patients will also receive a SDMG patient handout. The intervention addresses the previously identified challenges described above via an interactive and individualized electronic application designed to facilitate provision of SDMG.
  Arms: PAUSE App Intervention

SUMMARY:
Diabetes, heart disease and kidney disease have high morbidity and costs of care. Medications used to treat these conditions are effective. Yet, some have the risk of preventable adverse events when people are sick with the flu or stomach bug. These events include low blood sugar and acute kidney injury which can lead to extended hospital stays or death. Sick day medication guidance (SDMG) recommends stopping these medications temporarily when sick and restarted after symptoms subside. Unfortunately, many patients are not aware of these recommendations or find them hard to follow.

The investigator's previous research has shown that there is a lack of SDMG education and patient resources. Research on the development, implementation, usability and efficacy of these resources is also limited. In developing a SDMG tool, the investigators surveyed patients who expressed interest in an electronic health (eHealth) tool. As a result, the PAUSE App provides a timely and innovative way to provide continuity of care to patients that is linked to each patients' unique pharmacy record.

In the present pilot randomized control trial, the investigators will examine the outcomes of the PAUSE Initiative consisting of the PAUSE App and a SDMG educational handout. Approximately 16 Loblaw/Shoppers Drug Mart pharmacies across Alberta will take part. Patients of these pharmacies who take high-risk medications will be invited to participate. Each pharmacy will be randomized to provide their patients usual care (i.e. SDMG handout) or the intervention (i.e., PAUSE App + handout). Approximately 320 participants (20 per pharmacy) are expected to be recruited. The expected trial length is 9 months from recruitment to analysis.

A simulated 'sick day' survey will be used to assess the fidelity and efficacy of the PAUSE Initiative. Feasibility of the study processes (i.e., recruitment, onboarding) will be assessed to inform a full-scale trial. The usability and acceptability of the PAUSE App will also be investigated. Pharmacists and participants will complete questionnaires and qualitative interviews to assess these outcomes. Additionally, PAUSE App user metrics will be collected. All participants will receive an honorarium for their time.

DETAILED DESCRIPTION:
Our previous research surveyed healthcare providers from Alberta on "factors affecting clinician's decision to provide sick day medication guidance to patients with diabetes and CKD to prevent adverse events." Our results identified 75% of primary health providers were aware of sick day medication guidance, but just 56% knew where to find guidelines and resources. An overwhelming majority of respondents (97%) were supportive of enrolling patients in a study evaluating alternative innovations for providing sick day medication guidance.

In a recent scoping review summarizing existing interventions, our research team found the majority of published SDMG documents were aimed towards healthcare providers, with few patient-targeted documents. These were mainly in the form of handouts, wallet-sized cards, webpages, or telephone support. There is limited primary research on the development, implementation, or evaluation of current SDMG interventions. Most were reported to be challenging to follow and identification of sick days or qualifying medication without error was low. This survey and review highlight the need to develop and to evaluate new solutions for providing SDMG to patients. Our previous work also found that seniors in Canada were receptive to the use of electronic means of communication and several patients have expressed interest in using electronic health (eHealth) tools for sick day self-management.

Participants receiving the intervention will receive access to the PAUSE App, a self-management tool for SDMG intended for patients to use during an acute illness. Users' Loblaw/Shoppers Drug Mart pharmacy records are electronically linked to the PAUSE App within the President's Choice (PC) Health app allowing for up-to-date recommendations based on current prescribed medications. The app asks users a series of questions regarding signs and symptoms that identify a qualifying sick day illness, and screens for 'red flags' that would require emergency, or healthcare provider or urgent care referral, and help patients identify which of their medications they should temporarily withhold or adjusted, tailored to a patients' current medication list. This aims to provide patients with interactive support for managing medication during a sick day event. As part of the intervention, patients will also receive a SDMG patient handout. The intervention addresses the previously identified challenges of identifying qualifying signs and symptoms that warrant SDMG and which medications qualify via an interactive and individualized electronic application designed to facilitate provision of SDMG. The usual care group will receive a SDMG patient handout which outlines SDMG and addresses which medications qualify for SDMG.

Based on preliminary data, the investigators assume an absolute difference of 30% (50% with the PAUSE app vs. 20% without the PAUSE app) in the proportion of participants who complete a simulated sick day without error. Using a two-sided alpha of 0.05, 80% power, and an interclass correlation coefficient of 0.1 between pharmacy clusters, a sample size of 280 participants will be required. To account for a 10% loss to follow-up, the investigators will aim to recruit a total of 320 participants in the trial. The investigators plan to recruit 16 pharmacies that will recruit 20 participants each.

Data Analysis Participant baseline data, including sociodemographics, comorbidities, and active prescriptions will be analyzed using descriptive statistics. Feasibility and fidelity outcomes will be reported using descriptive statistics with numbers and percentages. Comparisons of outcomes between groups (e.g., PAUSE App vs. usual care) will be reported using unadjusted and adjusted generalized estimating equations to determine mean differences and risk differences between groups. Descriptive statistics will be used as appropriate to evaluate group differences following the follow-up period. Associations between key variables and study outcomes will be analyzed using appropriate univariate, multivariate, and mixed model analyses. Exploratory analyses of Google Analytics data will be performed to report user behaviour insights. Analyses of routinely collected health data over a 5-year extended follow-up period will be used to determine the effect, if any, of the intervention on health outcomes.

The simulated sick day evaluations will be scored and analyzed according to predefined scorecards based on scenarios used by Doerfler et al. measuring correct usage of SDMG during acute illness. Log-binomial regression models will be used to directly estimate the risk ratios (RRs) and 95% confidence intervals for the outcome of error free completion of the simulated sick day, as well as for correct completion of each of the 3 individual components of the sick day simulation. Random effects will be used to account for clustering by pharmacies. Unadjusted and adjusted models will be fit, including fixed effects for individual participant characteristics including age, sex, demographics, diabetes, other comorbidities, number of qualifying medications and any other significant confounding variables from univariate analyses. Additionally, data collected from participants on the usefulness of the PAUSE App and/or SDMG patient handout in managing a simulated sick day and overall acceptability of the interventions will be used to further assess the fidelity of the intervention. All statistical analysis will be completed in R.

Selected participants (patients and pharmacists) will be invited to be interviewed following their simulated sick day scenario evaluation based on the purposive sampling strategy. One-on-one semi-structured interviews will be conducted with participants and pharmacists ranging from 30-60 minutes in duration. Interview questions and analysis will be iterative throughout the study to allow for emerging or irregular themes to be examined in later interviews. Qualitative interviews will be audio-recorded, transcribed verbatim and examined using multiple phases of inductive thematic analysis. Collected field notes and transcriptions from interviews will be analyzed using NVIVO qualitative analysis software. Analysis of data will begin immediately following the conclusion of the first participant interview. Data will be coded by two researchers independently and then codes will be compared after the first interview to draft the coding manual for subsequent interviews.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age and able to provide informed consent
* be able to communicate (read, write, and speak) in English
* have access to a smartphone/tablet with an Internet connection
* be willing and able to download and use the PC Health app for the duration of the study
* currently be taking 2 or more medications from the following classes: renin-angiotensin-aldosterone system (RAAS) antagonists, diuretics, oral NSAIDs, metformin, or 1 or more medications from the following classes: insulin, sulfonylureas, meglitinides, SGLT2 inhibitors.

Exclusion Criteria:

* fail to meet the inclusion criteria
* have kidney failure requiring maintenance dialysis
* have had an organ transplant
* are pregnant
* receive qualifying medications in a blister pack or sachet
* do not primarily manage their own medications and condition (i.e., receive home care, in a rehabilitation or medical respite facility)
* cannot use the PC Health app independently
* previously participated in studies that led to the development of the PAUSE App (including the PAUSE study usability testing or needs assessment focus groups)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 3-month follow up
  Two to three patient participants on average per pharmacy per week can be recruited (320 patients from 16 pharmacies over 8 weeks)
Time to randomization | 3-month follow up
  ≥90% of study participants receive the intervention (SDMG handout, PAUSE App onboarding) to which they are randomized within 1 week of giving informed consent
Adherence to SDMG | 3-month follow up
  ≥50% of study participants randomized to pharmacies using the PAUSE app follow SDMG error-free during the simulated sick day evaluation.

SECONDARY OUTCOMES:
Exploration of participant experiences of study design and intervention acceptability | 3-month follow-up
  Semi-structured participant interviews will be undertaken to explore themes related to study design elements, such as pharmacist onboarding and education, and barriers and facilitators to understanding and usability of the PAUSE App intervention/SDMG tools. Coded concepts will be synthesized into overall themes inductively to form a comprehensive description of the data.
Exploration of pharmacist experiences of study design and intervention acceptability | 3-month follow-up
  Semi-structured pharmacist interviews will be undertaken to explore themes related to study design elements, such as onboarding procedures and education components, and experiences interacting with patients regarding the PAUSE App intervention and SDMG education. Coded concepts will be synthesized into overall themes inductively to form a comprehensive description of the data.
Exploration of PAUSE App-generated user behaviours and usage patterns | Throughout the 3-month data collection period
  Routinely collected, app-generated Google Analytics data will be captured over the data collection period to explore summary data trends, including but not limited to: total number of app visits, session duration, clicks on various pages within the app, time of day most frequently used, PDF (e.g., sick day guidance resources) downloads, and in-app engagement.
Exploration of the efficacy of the intervention in managing a simulated sick day event | At baseline and 3-month follow-up
  Pre- and post-intervention evaluation of paraticipant medication self-management using a 13-item Self-efficacy for Appropriate Medication Use Scale (SEAMS-13) survey.

OTHER OUTCOMES:
Exploration of future health outcomes summary data resultant of adverse drug-related events | Over an extended follow-up period of 5 years, or death (whichever comes first)
  Utilization of future health summary and administrative data to determine the difference, if any, of the intervention on all-cause health outcomes.
  Proposed collected summary data may include:
  * Increases in serum creatinine (mg/dl) based on the 2012 Kidney Disease Improving Global Outcomes (KDIGO) Clinical Practice Guidelines for AKI and AKD (i.e., >/= 0.3 mg/dl increase or 1.5-1.9x baseline serum creatinine)
  * Hospital admissions and emergency department data related to AKI and/or SDMG-related health outcomes
  * Vital statistics (e.g., death records) summary data related to AKI
  * Prescription medication history summary data related to AKI, worsening chronic conditions and/or SDMG

CONTACTS AND LOCATIONS:
Overall Officials: Ross T Tsuyuki, PharmD, Principal Investigator — University of Alberta; David JT Campbell, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Watson KE, Dhaliwal K, McMurtry E, Donald T, Lamont N, Benterud E, Kung JY, Robertshaw S, Verdin N, Drall KM, Donald M, Campbell DJT, McBrien K, Tsuyuki RT, Pannu N, James MT. Sick Day Medication Guidance for People With Diabetes, Kidney Disease, or Cardiovascular Disease: A Systematic Scoping Review. Kidney Med. 2022 May 28;4(9):100491. doi: 10.1016/j.xkme.2022.100491. eCollection 2022 Sep. PMID 36046611
- [Background] Watson KE, Dhaliwal K, Robertshaw S, Verdin N, Benterud E, Lamont N, Drall KM, McBrien K, Donald M, Tsuyuki RT, Campbell DJT, Pannu N, James MT; PAUSE (Preventing Medication Complications During Acute Illness Through Symptom Evaluation and Sick Day Guidance) Medication Safety Advisory Panel. Consensus Recommendations for Sick Day Medication Guidance for People With Diabetes, Kidney, or Cardiovascular Disease: A Modified Delphi Process. Am J Kidney Dis. 2023 May;81(5):564-574. doi: 10.1053/j.ajkd.2022.10.012. Epub 2022 Dec 5. PMID 36470530
- [Background] Dhaliwal KK, Watson KE, Lamont NC, Drall KM, Donald M, James MT, Robertshaw S, Verdin N, Benterud E, McBrien K, Gil S, Tsuyuki RT, Pannu N, Campbell DJT. Managing 'sick days' in patients with chronic conditions: An exploration of patient and healthcare provider experiences. Health Expect. 2023 Aug;26(4):1746-1756. doi: 10.1111/hex.13789. Epub 2023 Jun 8. PMID 37291977
- [Background] Watson KE, Dhaliwal K, Benterud E, Robertshaw S, Verdin N, McMurtry E, Lamont N, Drall KM, Gill S, Campbell DJT, McBrien K, Tsuyuki RT, Pannu N, James MT, Donald M. Managing Medications During "Sick Days" in Patients With Diabetes, Kidney, and Cardiovascular Conditions: A Theory-informed Approach to Intervention Design and Implementation. Can J Diabetes. 2024 Jun;48(4):259-268.e4. doi: 10.1016/j.jcjd.2024.02.003. Epub 2024 Feb 21. PMID 38395301